CLINICAL TRIAL: NCT02803983
Title: An Multicenter Prospective Observational Study to Pediatric Hip Plate Versus Cannulated Screw in Pediatric Femoral Neck Fracture (Delbet Type II and III)
Brief Title: Pediatric Hip Plate Versus Cannulated Screw in Pediatric Femoral Neck Fracture
Acronym: PFNF
Status: Completed | Type: Observational
Sponsor: The Fuzhou No 2 Hospital (Other)
Responsible Party: Principal Investigator, Shunyou Chen, Director,Orthopaedics, The Fuzhou No 2 Hospital
Other Study IDs: SChen
Record Dates: First submitted 2016-06-02; First posted 2016-06-17 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2016-06

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pediatric hip plate: The children were treated with pediatric hip plate.
  Interventions: Procedure: Pediatric hip plate
- Cannulated screw: The children were treated with cannulated screw.
  Interventions: Procedure: Cannulated screw

INTERVENTIONS:
Procedure: Pediatric hip plate — Children were treated with pediatric hip plate.
  Groups: Pediatric hip plate
Procedure: Cannulated screw — Children were treated with cannulated screw.
  Groups: Cannulated screw

SUMMARY:
The purpose of this study is to compare the early postoperative radiologic and clinical outcomes of pediatric hip plate and cannulated screw fixation in pediatric femoral neck fracture (Delbet type II and Delbet type III).

DETAILED DESCRIPTION:
The children aged 3 to 14 years with femoral neck fracture that were treated with pediatric hip plate and cannulated screw fixation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fractures that met these criteria, underwent definitive surgery and had complete clinical and radiographic follow up until fracture union at either institution were included in this study.

Exclusion Criteria:

* Pathologic fractures, and fractures in patients with osteogenesis imperfecta, neuromuscular disorders or any systemic disease that was associated with a predisposition to fractures or altered fracture healing were excluded.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric femoral neck fracture(Delbet type II and Delbet type III)
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Radiographic union | Through study completion, an average of 0.5 year.
  The time of radiographic union.

SECONDARY OUTCOMES:
The Ratliff classification standard score | Through study completion, an average of 1 year.
  Ratliff classification standard score was administered to determine the pain, function, activity and radiographic change.

OTHER OUTCOMES:
The complication | Through study completion, an average of 1 year.
  The complication was evaluated by osteonecrosis, epiphyseal arrest, premature physeal closure, limb length discrepancy (over 3 cm) and internal fixation failure.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] RATLIFF AH. Fractures of the neck of the femur in children. J Bone Joint Surg Br. 1962 Aug;44-B:528-42. doi: 10.1302/0301-620X.44B3.528. No abstract available. PMID 14038616
- [Result] Joeris A, Audige L, Ziebarth K, Slongo T. The Locking Compression Paediatric Hip Plate: technical guide and critical analysis. Int Orthop. 2012 Nov;36(11):2299-306. doi: 10.1007/s00264-012-1643-1. Epub 2012 Aug 26. PMID 22923267